CLINICAL TRIAL: NCT06083402
Title: Evaluating the Efficacy of a Dietary Supplement on Parameters of Skin Aging: a 12-Week, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Efficacy of a Dietary Supplement on Parameters of Skin Aging in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natals, Inc. dba Ritual (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HyaCera2023
Record Dates: First submitted 2023-08-16; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Skin Aging
Keywords: skin aging; skin wrinkles; skin hydration; skin elasticity; skin firmness; skin smoothness; crow's feet wrinkles; dietary supplement; skin barrier function

STUDY DESIGN:
Intervention Model Description: Healthy men and women with mild to moderate signs of skin aging will be randomly assigned to either receive a Ritual HyaCera or placebo for 12 weeks
Who Masked: Participant, Investigator
Masking Description: Neither the participants nor the investigators will know the group assignment. Supplements will be prepared by the sponsor and marked with unidentifiable ID numbers before being sent to study site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Participants receive 1 HyaCera™ capsule orally once daily for 12 weeks
  Interventions: Dietary Supplement: HyaCera™
- Placebo (Placebo Comparator): Participants receive 1 placebo capsule orally once daily for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HyaCera™ — 1 Ritual HyaCera capsule once daily
  Arms: Active
Dietary Supplement: Placebo — 1 placebo capsule once daily
  Arms: Placebo

SUMMARY:
As the body ages, the skin experiences natural changes in structure and composition. These changes may manifest visibly as increased skin dryness, wrinkling, and a loss of firmness/elasticity. In this double-blind, randomized, placebo-controlled trial, the investigators will recruit healthy men and women with mild to moderate signs of skin aging and randomly assign them to either receive a HyaCera™ or placebo for 12 weeks. The investigators will perform a series of objective and subjective measurements to assess changes in skin condition. The investigators hypothesize that consumption of HyaCera™ leads to improvements in the general condition of the skin including skin hydration, crow's feet wrinkling, and other skin aging parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 25 - 70 years old with mild to moderate fine lines and wrinkles
* All ethnicities and skin types
* Willing to maintain current skincare regimen on face, arms, and legs and withhold all facial and body treatments throughout the course of the study

Exclusion Criteria:

* Self-reported pregnant or breastfeeding or planning to become pregnant during the course of the study
* Any conditions on the face, arms and legs that would interfere with evaluations
* Under treatment for any known health issues/medical conditions including chronic health conditions and skin diseases/conditions

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Crow's Feet Wrinkles | at week 0, Week 4, Week 8, and Week 12
  Degree of crow's feet wrinkling will be measured via Visioscan®
Skin Smoothness | at week 0, Week 4, Week 8, and Week 12
  Skin smoothness will be measured via Visioscan®
Skin Hydration | at week 0, Week 4, Week 8, and Week 12
  Skin surface hydration will be measured via Corneometer® 825

SECONDARY OUTCOMES:
Skin Elasticity | at week 0, Week 4, Week 8, and Week 12
  Skin elasticity will be measured via Cutometer® MPA 580
Skin Barrier Function | at week 0, Week 4, Week 8, and Week 12
  Skin barrier function (as transepidermal water loss) will be measured via Tewameter®
Skin Scaliness | at week 0, Week 4, Week 8, and Week 12
  Skin scaliness will be measured via Visioscan®

OTHER OUTCOMES:
Dermatologist grading of skin condition | at week 0, Week 4, Week 8, and Week 12
  Visual and tactile dermatologist evaluation of skin condition (fine lines in the crow's feet area, wrinkles in the crow's feet area, skin dryness, skin radiance, and skin smoothness) based on 10-point grading scale (with 0 being no signs of aging and 9 being the most severe)
Self-evaluation of perceived changes in skin condition | at week 0, Week 4, Week 8, and Week 12
  Self-evaluation of changes in skin condition and signs of skin aging (i.e. fine lines & wrinkles, skin texture, skin smoothness, skin plumpness, skin glow/radiance, skin hydration, skin elasticity, skin redness, skin itchiness) using a 5-point Likert scale (options: much worse, somewhat worse, stayed the same, somewhat better, much better)

CONTACTS AND LOCATIONS:
Locations (1):
- Princeton Consumer Research, Raritan, New Jersey, United States

REFERENCES:
- [Derived] Grier-Welch AM, Vance AY, Alamdari N, Sharafi M. Efficacy of an Oral Skincare Supplement on Skin Aging: A 12-Week Randomized, Double-Blind, Placebo-Controlled Trial. Dermatol Ther (Heidelb). 2025 Dec;15(12):3689-3702. doi: 10.1007/s13555-025-01556-2. Epub 2025 Oct 10. PMID 41071523